CLINICAL TRIAL: NCT01310010
Title: Multicenter, Non-randomized Phase II Pilot Study to Assess the Efficacy and Safety of Dasatinib After Allogeneic Stem Cell Transplantation in Patients With de Novo Philadelphia Positive (Bcr-abl +) Acute Lymphoblastic Leukemia
Brief Title: Study of Dasatinib to Treat Philadelphia Positive Acute Lymphoblastic Leukemia
Acronym: DASA-TRAS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Grupo Espanol de trasplantes hematopoyeticos y terapia celular (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DASA-TRAS
Record Dates: First submitted 2011-02-10; First posted 2011-03-07 (Estimated); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: Leukemia, Lymphoblastic, Acute, Philadelphia-Positive
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Dasatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dasatinib (Experimental)
  Interventions: Drug: dasatinib

INTERVENTIONS:
Drug: dasatinib — Treatment with 100 mg QD of dasatinib (Sprycel®) administered orally as continuous daily dosing (CDD).
  Other Names: (Sprycel®)

SUMMARY:
Study hypothesis:

Treatment with dasatinib 100 mg QD is safe and efficacious when given to patients with Ph+ ALL in the post SCT setting.

DETAILED DESCRIPTION:
Participants - inclusion criteria

1. Adult patients ≥ 18 years.
2. Diagnostic confirmation of de novo Ph+ ALL.
3. Patients in first/second CR (assessed by cytology, karyotyping and/or FISH) at transplantation.
4. Patients with sustained hematologic and cytogenetic CR at the time of study entry.
5. Any modality of allogeneic SCT.
6. Patients are in days between 120 until 180 after allogeneic SCT with stable graft.
7. Ability to understand and voluntarily sign the informed consent form.
8. Women of childbearing potential (WOCBP) must be using an adequate method of contraception to avoid pregnancy and have a negative pregnancy test, a maximum of 48 hours prior to study drug start.

Participants - exclusion criteria:

1. Patients with ECOG 3-4 at study entry
2. Any of the following laboratory abnormalities:

   * Absolute neutrophil count < 1.5 x 109/l or platelets < 75 x 109/l
   * Serum creatinine > 2.0 mg/dl (177 mmol/l).
   * Serum glutamic oxalacetic transaminase (SGOT) or serum glutamate pyruvate transaminase (SGPT) > 5,0 x upper limit of normal (ULN).
   * Total bilirubin > 3 mg/dl.
3. Known HIV infection or any other uncontrolled infection at study entry
4. Known pleural effusion of any grade at study entry.
5. Morphologic or cytogenetic or molecular relapse at study entry
6. Evidence of digestive dysfunction that could prevent administration of study therapy
7. Prior therapy with dasatinib during >21 days
8. Other concurrent malignancy at study entry
9. Uncontrolled or significant cardiovascular disease, including myocardial infarction within 6 months, uncontrolled angina within 3 months, prolonged QT interval, congestive heart failure within 3 months and clinically significant ventricular arrhythmias
10. Any psychiatric condition that could prevent patient from signing the informed consent o could put the patient at an unacceptable risk in case of participating in the trial
11. Subjects enrolled in another clinical trial at study entry. If patients have received other investigational agent, a minimum of 30 days wash-out period must have elapsed.

Primary Outcome measures

The primary objective of this study is to assess the efficacy of dasatinib maintenance in terms of Disease Free Survival at 2 years in patients with Ph+ ALL who receive maintenance with dasatinib after allogeneic SCT.

Secondary Outcome measures

.To assess the efficacy of maintenance with dasatinib in terms of duration of hematologic, cytogenetic and molecular remission, Relapse rate at 2 years, survival at 2 years, overall DFS, and Overall Survival (OS).

·To assess the safety and tolerability of dasatinib maintenance regimen after allogeneic SCT

Regarding the secondary objective "To assess the safety and tolerability of dasatinib maintenance regimen after allogeneic SCT", such safety analysis includes the frequency of all adverse events and laboratory abnormalities as well as frequency of dose interruptions, dose reductions and treatment discontinuation for drug-related toxicity. Frequency tables will be reported using the "All treated subjects" dataset. Safety will be reported for all treated patients and assessed by baseline findings, AEs and SAEs (definition, pattern, seriousness and intensity according to NCI CTCAE v3.0, relationship with dasatinib and outcome). Hematologic toxicity will be analyzed separately.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients ≥ 18 years
2. Diagnostic confirmation of de novo Ph+ ALL
3. Patients in first/second CR (assessed by cytology, karyotyping and/or FISH) at transplantation
4. Patients with sustained hematologic and cytogenetic CR at the time of study entry
5. Any modality of allogeneic SCT
6. Patients are in days between 120 until 180 after allogeneic SCT with stable graft.
7. Ability to understand and voluntarily sign the informed consent form
8. Women of childbearing potential (WOCBP) must be using an adequate method of contraception to avoid pregnancy and have a negative pregnancy test, a maximum of 48 hours prior to study drug start

Exclusion Criteria:

1. Patients with ECOG 3-4 at study entry
2. Any of the following laboratory abnormalities:

   * Absolute neutrophil count < 1.5 x 109/l or platelets < 75 x 109/l
   * Serum creatinine > 2.0 mg/dl (177 mmol/l).
   * Serum glutamic oxalacetic transaminase (SGOT) or serum glutamate pyruvate transaminase (SGPT) > 5,0 x upper limit of normal (ULN).
   * Total bilirubin > 3 mg/dl.
3. Known HIV infection or any other uncontrolled infection at study entry
4. Known pleural effusion of any grade at study entry.
5. Morphologic or cytogenetic or molecular relapse at study entry
6. Evidence of digestive dysfunction that could prevent administration of study therapy
7. Prior therapy with dasatinib during >21 days
8. Other concurrent malignancy at study entry
9. Uncontrolled or significant cardiovascular disease, including myocardial infarction within 6 months, uncontrolled angina within 3 months, prolonged QT interval, congestive heart failure within 3 months and clinically significant ventricular arrhythmias
10. Any psychiatric condition that could prevent patient from signing the informed consent o could put the patient at an unacceptable risk in case of participating in the trial
11. Subjects enrolled in another clinical trial at study entry. If patients have received other investigational agent, a minimum of 30 days wash-out period must have elapsed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2010-04; Primary Completion 2015-10 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
The efficacy of dasatinib | at 2 years
  The primary objective of this study is to assess the efficacy of dasatinib maintenance in terms of Disease Free Survival at 2 years in patients with Ph+ ALL who receive maintenance with dasatinib after allogeneic SCT.

SECONDARY OUTCOMES:
To assess the efficacy of maintenance with dasatinib in terms of duration of hematologic, cytogenetic and molecular remission | at 2 years
  To assess the efficacy of maintenance with dasatinib in terms of duration of hematologic, cytogenetic and molecular remission, Relapse rate at 2 years, survival at 2 years, overall DFS, and Overall Survival (OS).
To assess the safety and tolerability of dasatinib maintenance regimen after allogeneic SCT | at 2 years
  To assess the safety and tolerability of dasatinib maintenance regimen after allogeneic SCT

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Sanz, Doctor, Principal Investigator — Hospital La Fe de Valencia
Locations (1):
- Hospital La Fe, Valencia, Spain